CLINICAL TRIAL: NCT02866760
Title: Helping In-patients to Quit Smoking by Understanding Their Risk Perception, Behavior, and Attitudes Related to Smoking
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Other Study IDs: In-patient
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Smoking
Keywords: Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims at understanding the needs and concerns of Chinese current smoking patients, including their risk perceptions, and the behavior, attitudes, and experiences related to smoking and smoking cessation. Specifically, how smokers overcome withdrawal symptoms and cigarette cravings, as a result of banning on smoking in hospitals, will be explored. In addition, whether smokers will stop, resume or continue smoking after hospitalization will be investigated.

DETAILED DESCRIPTION:
As about 400,000 hospitalizations are attributable to smoking annually in Hong Kong, it is an excellent "teachable moment" for healthcare professionals to help patients quit smoking. To our knowledge, this is the first study to investigate the needs and concerns of Chinese current smoking patients, including their risk perceptions, and the behavior, attitudes, and experiences related to smoking and smoking cessation. The findings of this study have important implications for research and clinical practice.

Understanding how hospitalized smokers perceive the risks of smoking, and their behaviour, attitudes, experiences related to smoking, as well as their view on hospital smoking cessation service are essential prerequisites for the design of an effective and appropriate smoking cessation intervention that can help patients achieve a greater level of smoking abstinence and a lower level of relapse. Moreover, the results of this study can guide the development of protocols and interventions that will demystify the misconceptions about smoking among hospitalized smokers, increase their perception of the risks of continued smoking and benefits of quitting. Additionally, it is crucial to motivate more healthcare professionals to assess health behaviors of hospitalized smokers and to implement evidence-based interventions to help them quit smoking. Most importantly, healthcare professionals should be offered relevant training so as to enhance their self-efficacy and confidence in promoting smoking cessation to patients.

The study consists of 2 phases. During phase 1, a purposive sample of 30 current adult smokers who admit to either medical or surgical units of one of the largest cute hospitals in Hong Kong will be invited to have a 60-minute semi-structured interview. The risk perceptions, and the behaviour, attitudes, and experiences related to smoking and smoking cessation amongst Chinese current smoking patients will be explored. Concerning phase 2, a convenience sample of 382 adult patients who are current smokers or ex-smokers in the three out-patient clinics will be invited to response to the questionnaires. Based on the findings of Phase 1 study, a survey study will be conducted to further explore the behaviour, attitudes, and experiences related to smoking and smoking cessation amongst those patient who smoked before their admission to hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or above
2. able to speak Cantonese Phase 1:(3) current smokers, either occasional or daily(4) hospitalized for at least 48 hours Phase 2:(3) current smokers who have resumed smoking or ex-smokers who have quitted smoking after hospitalization(4) admitted to hospitals, either medical or surgical units during the past 3 months.

Exclusion Criteria:

1. unstable medical conditions, as advised by the doctor in charge
2. poor cognitive state or active psychotic symptoms

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase 1 Qualitative study:
  Chinese patients admitting to either medical or surgical units of one of the largest acute hospital in Hong Kong for physical discomfort.
  Phase 2 Survey study:
  Chinese patients attending one of the three general outpatient clinics at different regions in Hong Kong for medical follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2016-07; Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
The behavior, attitudes, and experiences related to smoking and smoking cessation among Chinese current smoking patients | 3 months
  1. smoking patients' risk perceptions, and the behavior, attitudes, and experiences related to smoking and smoking cessation
  2. how they overcome withdrawal symptoms and cigarette cravings, as well as their view on hospital smoking cessation service

SECONDARY OUTCOMES:
The behavior, attitudes, and experiences related to smoking and smoking cessation among those patients who smoked before their admission to hospitals | 10 months
  whether they (1) experience withdrawal symptoms or cigarette cravings and depressive symptoms during and after hospitalization (2)receive medical advice for quitting during hospitalization (3) have stopped, resumed or continued smoking after hospitalization (4) have intention to quit (5) have an increase in the risk perception toward smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho KY, Li WHC, Lam KKW, Wang MP, Xia W, Ho LY, Tan KCB, Sin HKM, Cheung E, Mok MPH, Lam TH. Smoking behaviours of Hong Kong Chinese hospitalised patients and predictors of smoking abstinence after discharge: a cross-sectional study. BMJ Open. 2018 Dec 19;8(12):e023965. doi: 10.1136/bmjopen-2018-023965. PMID 30573486